CLINICAL TRIAL: NCT02857842
Title: The Effect of Reduced Corticosteroid Therapy in Patients With Acute Exacerbation of COPD
Brief Title: Corticosteroid Reduction in COPD
Acronym: Cortico-cop
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Principal Investigator, Pradeesh Sivapalan, MD, Ph.d.-student, Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol_CORTICO-COP_PSJUJ
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Lung Diseases, Obstructive; Blood Eosinophil Count; Glucocorticoids; COPD; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blood eosinophil guided prednisolone treatment (Experimental): Intravenous Solu-Medrol 80 mg, followed by prednisolone tablet 37.5 mg daily (maximum of 5 days in all) if the eosinophil count in the blood ≥ 0.3 x 10E9/L. Eosinophil count in the blood <0.3 x 10E9/L results in no treatment with prednisolone. If the patient is discharged during the treatment period, given treatment from the last measured eosinophil count the remaining days.
  Interventions: Drug: Prednisolone
- Standard of care (Active Comparator): Intravenous Solu-Medrol 80 mg on the first day followed by 37.5 mg of prednisolone tablets (1 x 25 mg plus 1 x 12.5 mg) daily for 5 days
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone

SUMMARY:
This study explores whether patients hospitalized with chronic obstructive pulmonary disease (COPD) exacerbation may have fewer days with prednisolone and with the same treatment effect by controlling the treatment by daily measurements of eosinophils.

DETAILED DESCRIPTION:
The most commonly used treatment for acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is a 5-day treatment with corticosteroids in moderate-high dose. Some patients receive repeated treatments, although it has been shown that corticosteroids only have temporary beneficial effects and no effect in relation to serious incidents or mortality. It has been found that the higher accumulated prednisolone dose disables patients due to serious side effects, including pneumonia, dysregulated diabetes, bone fracture in the context of osteoporosis, mental disorder and adrenal insufficiency etc. However, the extent of the side effects is unknown. Recent research has shown that it is presumably only a small subset of COPD patients who benefit from corticosteroid therapy. This group can be identified by the biomarker "blood-eosinophils" as already measured on most AECOPD patients during hospitalization.

This is a randomized, controlled, multi-center, non-Inferiority trial evaluating the effect of eosinophil guided corticosteroid therapy to patients with AECOPD. The aim of the study is to investigate whether the accumulated dose corticosteroid treatment during admissions for AECOPD can be reduced, including the presumed side effects, while (still) remaining the optimal treatment effect.

ELIGIBILITY:
Inclusion criteria:

* Patients hospitalized with AECOPD
* Age ≥ 40 years
* Spirometry-verified COPD (defined as FEV1 / FVC ≤ 70%)
* Chronic Obstructive Lung Disease (GOLD) class C or D
* Inclusion within 24 hours after admission

Exclusion criteria:

* Known with a diagnosis of asthma
* Life expectancy less than 30 days
* Serious exacerbation requiring invasive ventilation or admission to ICU
* Allergy to systemic corticosteroids
* Severe mental illness, which is not controlled by medication
* People who are detained under the act on the use of coercion in psychiatry
* Severe language problems or inability to provide written informed consent
* Pregnancy and lactation
* Systemic fungal infections

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2016-08; Primary Completion 2018-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Days alive and out of hospital within 14 days after recruitment | 14 days from recruitment

SECONDARY OUTCOMES:
Treatment failure (Recurrence of AECOPD resulting in emergency room visits, hospitalization or need to intensify pharmacological treatment within 30 days) | 30 days
Change in lung function (ΔFEV1) on day 3, after 1 month and 3 month | 90 days
Mortality | 360 days
Infection requiring antibiotic treatment within 180 days after the index of AECOPD | 180 days
The period between index AECOPD and the next AECOPD exacerbation | 90 days
  1. Readmission with AECOPD or death
  2. Time to readmission with AECOPD or death
Cumulative corticosteroid dose at 1 and 3 month follow-up | 90 days
  1. Proportions of patients using corticosteroids during hospitalization (day 1 to day 5) between treatment arms
  2. Mean total cumulative dose from recruitment to 3-month follow-up
Hyperglycemia during admission | 14 days
Changes in PTH and Vitamin D status between hospitalization and 3-month follow-up | 90 days
Change in bone marker levels (Serum P1NP, Serum CTX) | 90 days
Dyspepsia or ulcer complications (gastrointestinal bleeding) | 90 days
New onset or worsening of diabetes mellitus | 30 days
Increase in body mass index between hospitalization, at 30 days and 3-month follow-up | 90 days
The impact of COPD (cough, sputum, dysnea, chest tightsenes etc) on health status (COPD Assessment Test) between hospitalization, at 30 days and 3-month follow-up | 90 days
Changes in level of dyspnea using the Medical Research Council (MRC) Dyspnoea Scale between hospitalization, at 30 days and 3-month follow-up | 90 days
Osteoporotic fractures | 360 days

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Bispebjerg University Hospital, Copenhagen
  - Hvidovre University Hospital, Copenhagen
  - North Zealand Hospital, Copenhagen
  - Gentofte University Hospital, Hellerup

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Sivapalan P, Jorgensen NR, Mathioudakis AG, Eklof J, Lapperre T, Ulrik CS, Andreassen HF, Armbruster K, Sivapalan P, Janner J, Godtfredsen N, Weinreich UM, Nielsen TL, Seersholm N, Wilcke T, Schuetz P, Klausen TW, Marsa K, Vestbo J, Jensen JU. Bone turnover biomarkers in COPD patients randomized to either a regular or shortened course of corticosteroids: a substudy of the randomized controlled CORTICO-COP trial. Respir Res. 2020 Oct 12;21(1):263. doi: 10.1186/s12931-020-01531-9. PMID 33046053
- [Derived] Sivapalan P, Lapperre TS, Janner J, Laub RR, Moberg M, Bech CS, Eklof J, Holm FS, Armbruster K, Sivapalan P, Mosbech C, Ali AKM, Seersholm N, Wilcke JT, Brondum E, Sonne TP, Ronholt F, Andreassen HF, Ulrik CS, Vestbo J, Jensen JS. Eosinophil-guided corticosteroid therapy in patients admitted to hospital with COPD exacerbation (CORTICO-COP): a multicentre, randomised, controlled, open-label, non-inferiority trial. Lancet Respir Med. 2019 Aug;7(8):699-709. doi: 10.1016/S2213-2600(19)30176-6. Epub 2019 May 20. PMID 31122894
- [Derived] Sivapalan P, Moberg M, Eklof J, Janner J, Vestbo J, Laub RR, Browatzki A, Armbruster K, Wilcke JT, Seersholm N, Weinreich UM, Titlestad IL, Andreassen HF, Ulrik CS, Bodtger U, Nielsen TL, Hansen EF, Jensen JUS. A multi-center randomized, controlled, open-label trial evaluating the effects of eosinophil-guided corticosteroid-sparing therapy in hospitalised patients with COPD exacerbations - The CORTICO steroid reduction in COPD (CORTICO-COP) study protocol. BMC Pulm Med. 2017 Aug 15;17(1):114. doi: 10.1186/s12890-017-0458-7. PMID 28810909
- See also: Related Info — http://www.coptrin.dk